CLINICAL TRIAL: NCT04230031
Title: LCI-HEM-MYE-PurD-001: Phase II Study of Daratumumab Pre-Mobilization and Post-Autologous Stem Cell Transplant in Patients With Multiple Myeloma and Sub-Optimal Response to Induction
Brief Title: Phase II Study of Daratumumab Pre-Mobilization and Post-ASCT in Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult enrollment due to changes in standard of care
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-HEM-MYE-PURD-001; 00040671 (Other: Advarra IRB)
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1: Daratumumab (Experimental): Pre-ASCT and Post-ASCT: Daratumumab
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Experimental
  Other Names: Darzalex

SUMMARY:
This study will use the drug daratumumab in patients who did not achieve at least a very good partial response (VGPR) and are already planned to have an Autologous Stem Cell Transplant (ASCT). Daratumumab will be given before the stem cell collection to attempt to get rid of any multiple myeloma cells that may be present in the stem cell collection and after the ASCT to get rid of any multiple myeloma cells that may be remaining.

DETAILED DESCRIPTION:
This is a single arm, two-stage, phase II study to evaluate the rate of ≥ Complete Response (CR) post-Autologous Stem Cell Transplant (ASCT) in Multiple Myeloma (MM) subjects who failed to achieve at least a Very Good Partial Response (VGPR) post initial induction therapy for newly diagnosed disease, and for whom an ASCT is planned. Subjects will be treated with four weekly doses of daratumumab before mobilization for Hematopoietic Progenitor Cells (HPC) collection, followed by high dose chemotherapy and ASCT and four weekly doses of daratumumab after ASCT. A two-stage design will be implemented. Twenty three (23) subjects will be enrolled in the first stage, and if at least 12 of the 23 subjects have at least a CR after ASCT, an additional 16 subjects will be enrolled in the second stage (a total of 39 subjects).

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. ≥ 18 years of age
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 within 28 days prior to day 1 of daratumumab.
4. Failure to achieve a VGPR or better per IMWG 2016 criteria following a three-drug induction regimen for newly diagnosed MM. Subjects must have achieved at least minimal response to induction therapy.
5. Measurable disease at time of diagnosis (collected within 42 days prior to initiation of initial induction therapy) defined as:

   1. Serum M-protein ≥ 0.5. g/dL OR
   2. Urine M-protein ≥ 200 mg/24 h OR
   3. Involved free light chain (FLC) level ≥ 10 mg/dL provided serum FLC ratio is abnormal
6. ASCT is planned for post-induction therapy.
7. Prior radiotherapy must be completed at least 14 days prior to day 1 of daratumumab and subject must have recovered from any radiation-induced toxicities.
8. Recovered from all reversible acute toxic effects of induction therapy (other than alopecia) to ≤Grade 1 or baseline.
9. Demonstrate adequate organ function within 28 days of day 1 of daratumumab as defined in the table below:

   * White Blood Cell (WBC) ≥ 2,000/mm3
   * Absolute Neutrophil Count (ANC) ≥ 1,000/mm3 without growth factors for 1 week prior
   * Hemoglobin (Hgb) ≥ 8 g/dL
   * Platelet count ≥ 70,000/mm3 if bone marrow plasmacytosis of <50%; otherwise ≥ 50,000/mm3(*)
   * Serum creatinine OR Creatinine clearance ≤ 1.5 × upper limit of normal (ULN) OR ≥ 30 mL/min as measured by a 24-hour urine collection or estimated by the Cockcroft - Gault formula
   * Bilirubin ≤ 2 × ULN; < 3.0 for subjects with Gilbert's Syndrome
   * Aspartate aminotransferase (AST) ≤ 2.5× ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
10. Females of childbearing potential (FCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to day 1 of daratumumab. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
11. FCBP must be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 90 days (3 months) after the last dose of daratumumab. Contraceptive methods with low user dependency are preferable but not required.
12. Male subjects who are sexually active with a FCBP must be willing to use condoms from the time of informed consent until 3 months after the last dose of daratumumab has been discontinued. The FCBP partner should also consider contraception recommendations (see inclusion #11).
13. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Active infection requiring systemic therapy (i.e., involving IV antibiotics)
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study, and any female subject must agree not to donate eggs during the study and for 3 months after the last dose of daratumumab).
3. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, carcinoma of the prostate with a current PSA value of <0.5 ng/mL or other cancer for which the subject has completed treatment, been disease-free for at least five years, and is considered by Sponsor-Investigator to be at <30% risk of relapse, or on hormonal therapy for a history of either prostate cancer or breast cancer, provided that there has been no evidence of disease progression during the previous three years.
4. Non-secretory MM.
5. Active involvement of the central nervous system by MM.
6. Prior cerebrovascular accident with persistent neurological deficit.
7. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
8. Had major surgery within 2 weeks prior to day 1 of daratumumab.
9. Treatment with any investigational drug within 4 weeks prior to day 1 of daratumumab.
10. Uncontrolled clinically significant illness including, but not limited to, uncontrolled hypertension (as per the most updated Joint National Committee for the Management of Hypertension definitions), symptomatic congestive heart failure (as per New York Heart Association [NYHA] class III or IV [see Appendix C], uncontrolled angina pectoris, myocardial infarction within the past 6 months from consent, known or suspected amyloidosis, uncontrolled cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator, or any other condition (including laboratory abnormalities) that would, in the opinion of the Sponsor-Investigator, place the subject at unacceptable risk if he/she were to participate in the study.
11. Known allergies, hypersensitivity or intolerance to monoclonal antibodies or human proteins, daratumumab or its excipients.
12. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
13. Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
14. Is known to be seropositive for human immunodeficiency virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate Post-ASCT | up to 100 days post-ASCT
  CR or better will be determined for each subject as binary variables indicating whether or not best overall response post-ASCT is a CR or better as determined by the IMWG 2016 response criteria.

SECONDARY OUTCOMES:
VGPR+ Rate | up to 100 days post-ASCT
  Post ASCT VGPR+ response will be determined for each subject as a binary variable indicating whether or not the subject achieved a post-ASCT response of VGPR or better as determined by the IMWG response criteria
Time to First Response (TTFR) | up to 100 days post-ASCT
  TTFR is defined as the time from start of induction therapy to the time when the first occurrence of a post-ASCT VGPR or better was achieved.
Time to Best Response (TTBR) | up to 100 days post-ASCT
  TTBR is defined as the time from start of induction therapy to the time when the best response of VGPR or better was achieved.
Duration of Response (DOR) | up to 7 years
  DoR will be calculated separately for each subject achieving PR or better, VGPR or better, and CR or better. The DoR intervals will be calculated from the time of the first assessment that identified response until disease progression or death from any cause.
Progression-Free Survival (PFS) | up to 7 years
  PFS is defined as the duration of time from start of induction therapy to first occurrence of either progressive disease or death from any cause
Time to Progression (TTP) | up to 7 years
  TTP will be calculated in the same fashion as described for PFS with the exception that for subjects who die for causes other than disease progression.
Time to Next Treatment (TTNT) | up to 7 years
  TTNT will be calculated from start of induction therapy until the start of the first subsequent anti-cancer therapy after all protocol directed therapy is completed.
Overall Survival (OS) | up to 7 years
  OS is defined as the duration from start of induction therapy to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shebli Atrash, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided